CLINICAL TRIAL: NCT00645775
Title: The Efficacy of Irvingia Gabonensis (Bush Mango) in the Management of Overweight, Obesity and Metabolic Syndrome in Cameroon.
Brief Title: Effect of Irvingia Gabonensis (Bush Mango)on Parameters Associated With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gateway Health Alliance (Industry)
Collaborators: University of Yaounde (Other)
Responsible Party: Pr. Julius Oben, CSO, Gateway Health Alliances
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GHAIGOB131CT
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2006-08

CONDITIONS: Metabolic Syndrome; Obesity; Dyslipidemia
Keywords: Weight loss; Antiobesity; Metabolic syndrome; Leptin
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Dyslipidemias; Weight Loss | interventions — IGOB131

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Placebo Comparator): Compare active to placebo
  Interventions: Dietary Supplement: IGOB131

INTERVENTIONS:
Dietary Supplement: IGOB131 — Comparison of 250 mg per day of Irvingia gabonensis to placebo

SUMMARY:
The study investigated the use and efficacy of the seeds of African bush mango (Irvingia gabonensis)to control body weight, blood lipids and hormones in overweight and obese people.

DETAILED DESCRIPTION:
To assess the effects of seeds of Irvingia gabonensis on body weight, fasting blood glucose, plasma total and LDL cholesterol in 102 overweight and obese participants.

The study was a 10 week randomized, double blind, placebo controlled design. participants were randomly divided into 2 groups of 51 participants each. Group 1 was the placebo group, while Group 2 was the active group. Each group received 2 daily doses of 125 mg (before meals) of either placebo or Irvingia gabonensis.

Weight as well as fasting blood was taken at baseline and at 4, 8 and 10 weeks. No major detary changes or exercises were suggested during the study period.

ELIGIBILITY:
Inclusion Criteria:

* BMI>26

Exclusion Criteria:

* Diabetics Pregnant and lactating Participating in any other weight reducing program Smokers

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2006-11; Primary Completion 2007-03 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Weight change | 10 weeks

SECONDARY OUTCOMES:
Change in blood lipids and hormone levels | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Julius E Oben, PhD, Study Director — Gateway Health Alliances / University of Yaounde
Locations (1):
- Laboratory of Nutrition & Nutritional Biochemistry, Yaoundé, Centre Region, Cameroon

REFERENCES:
- [Derived] Ngondi JL, Etoundi BC, Nyangono CB, Mbofung CM, Oben JE. IGOB131, a novel seed extract of the West African plant Irvingia gabonensis, significantly reduces body weight and improves metabolic parameters in overweight humans in a randomized double-blind placebo controlled investigation. Lipids Health Dis. 2009 Mar 2;8:7. doi: 10.1186/1476-511X-8-7. PMID 19254366